CLINICAL TRIAL: NCT01050582
Title: Evaluation of Growth, Sexual Maturation, and Prolactin-Related Adverse Events in the Pediatric Population Exposed to Atypical Antipsychotic Drugs
Brief Title: A Study to Evaluate the Safety and the Effects of Risperidone Compared With Other Atypical Antipsychotic Drugs on the Growth and Sexual Maturation in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR016687; RISNAP4022 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Results first posted 2012-11-27 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-10

CONDITIONS: Schizophrenia; Bipolar Disorder; Autistic Disorder; Conduct and Other Disruptive Behavior Disorders
Keywords: Schizophrenia; Bipolar Disorder; Autistic Disorder; Conduct and Other Disruptive Behavior Disorders; Risperidone; RISPERDAL; Antipsychotic Agents; Prolactin; Pediatrics
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Autistic Disorder; Behavior | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risperidone (Experimental): Risperidone as per local prescribing practices
  Interventions: Drug: Risperidone
- Other atypical antipsychotic drugs (Experimental): Other atypical antipsychotic drugs as per local prescribing practices
  Interventions: Drug: Other atypical antipsychotic drugs

INTERVENTIONS:
Drug: Risperidone — As per local prescribing practices
  Arms: Risperidone
Drug: Other atypical antipsychotic drugs — As per local prescribing practices
  Arms: Other atypical antipsychotic drugs

SUMMARY:
The purpose of this study is to evaluate the effects of risperidone compared with other atypical antipsychotic drugs on the physical maturity, growth and development of children, and the risk of prolactin-related adverse events (side effects) associated to these drugs.

DETAILED DESCRIPTION:
This is a study to find out what the effects are of long-term use of atypical antipsychotics (drugs used to treat mental health and some behavior disorders) in children and adolescents on their growth and physical maturity. Atypical antipsychotics are used in the treatment of a wide range of disorders in children and adolescents, such as; schizophrenia, bipolar mania, autistic disorder or other disruptive behavior disorders. This study does not involve using any new medication, but to look into some of the side effects that children and adolescents may experience from taking an atypical antipsychotic. One of the side effects of some atypical antipsychotics is an increased level of "prolactin", a hormone that occurs naturally in the body which can lead to "hyperprolactinemia" a condition in which the pituitary gland produces too much prolactin. In order to further investigate these possible side effects, two groups of children and adolescents (aged 8 to 16) with a diagnosis of schizophrenia, bipolar mania, autistic disorder, or conduct and other disruptive behavior disorders who are or have been recently treated with an atypical antipsychotic will be enrolled; 1 group of children and adolescents will either be currently taking or have recently been treated with risperidone and the second group of children and adolescents will either be currently taking or have recently been treated with an a similar type of atypical antipsychotic therapy. The results will then be compared to see if the age of physical maturation, growth and development differs between the two groups, using data collected during an office visit and previous information available from existing medical records. The patient's growth will be assessed using information on height and weight taken from the medical records at different time points before (up to one year previous) and since they started treatment with antipsychotic therapy. In addition, there will also be one visit to the clinic where the growth and stage of sexual maturity of the patient will be reviewed by both the study doctor and through the patient's own assessment, using a questionnaire and pictures developed specially to assess stages of physical development (so called - Tanner stage). In addition, one blood sample will be taken from each patient to check the levels of prolactin hormone in the blood to see if this differs between treatment groups. Potential patients will be identified through automated databases and/or medical chart review. If, after fully understanding the purpose of this study, the parent, legal guardian and their child agree to participate by signing an informed consent (children to sign an assent form), information (specified below) related to your child's treatment and development will be collected directly from central medical records or from notes kept by your child's doctor for evaluation. The following data will be collected from available medical records: information about the patient's use of antipsychotic drug and prescriptions; previous records of the patient's height, weight, and growth; physical and sexual development (so called, Tanner stage [developmental stage]) if available; results of previous blood tests taken to evaluate the level of the hormone prolactin if available; and, history of any side effects that could be related to increased levels of the hormone prolactin. All the above information will be collected within 1 year before the patient started antipsychotic therapy. The same information (if available) will also be collected following the time that the patient starting taking their atypical antipsychotic medication until the present time. As much information as possible will be collected for this period of time so that a determination of how taking antipsychotic drugs may have influenced the patient's growth can be made. The study doctor will see each patient for a single study visit. This visit will take place at a convenient time approximately one week after informed consent/assent has been obtained. At the clinic visit, the study doctor will do some examinations to check the patient's general health and assess their growth and physical development. These will include: a physical examination (including developmental stage assessment [Tanner stage]), weight and height, vital signs (pulse, respiration rate, temperature and blood pressure), medical history, and the collection of information regarding the occurrence of any side effects thought to be related to the use of atypical antipsychotic medication or related to the hormone prolactin. In addition to being assessed by the study doctor, the patient will be asked to complete the Tanner Stage questionnaire. This will involve the patient reviewing both pictures and written descriptions of children at different stages of physical development. The patient will have to decide which picture/description is most representative of their body. The study doctor will also look at the patient's current use of any other medications. Each patient will participate in the study for about one week. The outcome measures of the study will be to compare Z-scores for height, age at current Tanner stage, and prolactin-related adverse events between patients exposed to risperidone and patients exposed to other atypical antipsychotic drugs. Outcome measures will be collected during the study visit and retrospectively during the time of exposure for up to 2 years prior to the study visit.

ELIGIBILITY:
Inclusion Criteria:

* One or both parents (according to local regulations) or a guardian must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study (If appropriate according to local regulations, the patient must also assent)
* Treated for schizophrenia, bipolar mania, autistic disorder, or conduct and other disruptive behavior disorders
* Had at least 6 months of exposure for an atypical antipsychotic drug within 24 months before the study visit (patients may or may not be taking the atypical antipsychotics at the time of actual enrollment, eligible patients can have exposure to multiple atypical antipsychotics, however, they cannot concomitantly be exposed to more than 1 atypical antipsychotic for a period of greater than 30 days)
* Had medical records or automated data available for at least 1 year prior to the start of exposure
* Height and weight were recorded at least once within 1 year before the start of exposure, and if available at any time points after the start of exposure in the medical records or electronic databases (not mandatory)

Exclusion Criteria:

* Have at least 1 medical record, at any time before the start of exposure, consistent with malignancy (other than non-melanoma skin cancer), pregnancy, or a developmental delay or abnormality associated with growth or sexual maturation delays not related to the specified indications
* Had exposure to prolactin elevating medications other than atypical antipsychotics and selective serotonin reuptake inhibitors (SSRIs)
* Had exposure to Paliperidone
* Cannot comply with study procedures

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 244 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (28):
- United States (13):
  - San Francisco, California
  - Aurora, Colorado
  - Altamonte Springs, Florida
  - Gainesville, Florida
  - Smyrna, Georgia
  - Naperville, Illinois
  - Indianapolis, Indiana
  - Valparaiso, Indiana
  - Boston, Massachusetts
  - Cambridge, Massachusetts
  - Glen Oaks, New York
  - Cleveland, Ohio
  - Columbus, Ohio
- Antwerp, Belgium
- Germany (7):
  - Freiburg im Breisgau
  - Jena
  - Mannheim
  - München
  - Tübingen
  - Ulm
  - Würzburg
- Athens, Greece
- Nijmegen, Netherlands
- Poland (5):
  - Gdansk
  - Kielce
  - Lódź
  - Sosnowiec
  - Warsaw

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 244 subjects were assessed for eligibility of whom 230 signed informed consent. Of the 230, 43 were found not to meet inclusion or exclusion criteria, 2 withdrew consent, and 1 was not kept in the study due to a site decision. A total of 184 subjects were included in the analysis.
Groups:
- Risperidone: Subjects with at least 6 months exposure to risperidone within 24 months prior to enrollment
- Other Atypical Antipsychotics: No risperidone exposure within 24 months of enrollment, no more than 30 days lifetime exposure to risperidone, and at least 6 months exposure to another atypical antipsychotic within 24 months prior to enrollment
Period: Overall Study
Arm/Group | Risperidone | Other Atypical Antipsychotics
Started | 133 | 51
Completed | 133 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risperidone | Other Atypical Antipsychotics | Total
Number analyzed (Participants) | 133 | 51 | 184
Age Continuous [Mean (Standard Deviation); unit: years] | 12 (2.5) | 12 (2.5) | 12 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 117 | 33 | 150
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 6 | 18
  White | 110 | 36 | 146
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 59 | 40 | 99
  Germany | 41 | 6 | 47
  Poland | 19 | 3 | 22
  Netherlands | 8 | 0 | 8
  Greece | 3 | 2 | 5
  Belgium | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Height (cm) Z-score at Study Visit
Description: Height (cm) measured at the study visit was converted to a Z-score based on the US Center for Disease Control 2000 growth charts for US subjects and European growth charts for ex-US subjects. A z-score indicates how many standard deviations a subject is away from the expected height for the subject's age and gender.
Time Frame: One single study visit, approximately one week after informed consent has been obtained
Population: All participants with a height assessment available at the study visit.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Risperidone | Other Atypical Antipsychotics
Number analyzed (Participants) | 132 | 50
z-score | 0.40 (1.189) | 0.09 (1.079)
Statistical Analysis 1: Comparison: Risperidone vs Other Atypical Antipsychotics; Null hypothesis is that there is no difference between the risperidone and other atypical antipsychotics groups in current height z-score; Test type: Superiority or Other; p < 0.001, Regression, Linear; Covariates: weight (wt) divided expected wt for age and height (ht), age, use of concomitant medication with growth effects, preexposure ht z-score; Slope = 0.447, 95% CI 2-sided [0.220 to 0.674], Standard Error of Mean 0.116 — Slope associated with treatment dummy variable with 1 indicating risperidone and 0 indicating other atypical antipychotics

2. Secondary Outcome: Age (Years) at Current Tanner Stage
Description: Tanner stage is an evaluation of pubertal development with values ranging from 1 (pre-pubertal) to 5 (adult). A standardized, validated tool containing standardized pictures and written descriptions of the stages of pubic hair development, breast development for girls, and genital development for boys was used by physicians to make their assessment.
Time Frame: One single study visit, approximately one week after informed consent has been obtained
Population: Participants with a physician assessed Tanner stage value.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Risperidone | Other Atypical Antipsychotics
Number analyzed (Participants) | 124 | 49
years
  Tanner Stage 1 | 10.2 (1.31) | 10.3 (1.78)
  Tanner Stage 2 | 11.3 (1.68) | 11.2 (1.73)
  Tanner Stage 3 | 13.1 (2.18) | 12.2 (1.21)
  Tanner Stage 4 | 14.9 (1.27) | 15.0 (1.46)
  Tanner Stage 5 | 15.1 (0.69) | 15.0 (1.82)
Statistical Analysis 1: Comparison: Risperidone vs Other Atypical Antipsychotics; The null hypothesis is that there is no difference between the risperidone and other atypical antipsychotics groups in age (years) at current Tanner stage; Test type: Superiority or Other; p = 0.378, Regression, Linear; Covariates: Tanner stage and gender; Slope = -0.221, 95% CI 2-sided [-0.711 to 0.269], Standard Error of Mean 0.250 — Slope associated with treatment dummy variable with 1 indicating risperidone and 0 indicating other atypical antipsychotics

3. Secondary Outcome: Number of Participants With Retrospectively Reported Potentially Prolactin-Related Adverse Events
Description: Previous potentially prolactin-related adverse events, including hyperprolactinemia, were reviewed and abstracted from participants' medical records. Potentially prolactin-related adverse events include breast symptoms, menstrual disorders, hyperprolactinemia, and prolactinoma.
Time Frame: Retrospectively during the time of exposure for up to 2 years prior to the study visit
Measure: Number; unit: participants
Arm/Group | Risperidone | Other Atypical Antipsychotics
Number analyzed (Participants) | 133 | 51
participants | 7 | 3
Statistical Analysis 1: Comparison: Risperidone vs Other Atypical Antipsychotics; Null hypothesis is that there is no difference between the risperidone and other atypical antipsychotics groups in frequency of retrospectively reported potentially prolactin-related adverse events; Test type: Superiority or Other; p > 0.999, Fisher Exact; Odds Ratio (OR) = 0.865, 95% CI [0.189 to 3.963] — Estimated OR is from a logistic regression model including factors for treatment arm, age, indication, and use of concomitant medication with growth effects

ADVERSE EVENTS:
Time Frame: Days from signing of informed consent to study visit
Description: Adverse events prospectively reported from the time of signing informed consent to the study visit are summarized.
Arm/Group | Risperidone | Other Atypical Antipsychotics
Serious Adverse Events (participants affected / at risk) | 0/133 | 0/51
Other Adverse Events (participants affected / at risk) | 8/133 | 3/51
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone (N=133) | Other Atypical Antipsychotics (N=51)
Blood prolactin increased (Investigations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Sedation (Nervous system disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Middle insomnia (Psychiatric disorders) | 1 | 0
Weight increased (Investigations) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Drug ineffective (General disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0
Oedema (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
A total of 350 subjects in a 1:1 ratio between the two arms was planned. Recruitment difficulties led to an imbalance in the number of subjects per arm and to early termination of the study. The results should be interpreted within this context.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No